CLINICAL TRIAL: NCT03863626
Title: Exploring Diuretics Effective Management in Acute Decompensated Heart Failure, EDEMA Trial
Acronym: EDEMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Collaborators: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmad Samir, Lecturer of Cardiovascular Medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-166-2018
Record Dates: First submitted 2019-02-23; First posted 2019-03-05 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Acute Decompensated Heart Failure; Diuretics Resistance

STUDY DESIGN:
Intervention Model Description: randomized controlled trial 2 equal groups for IV shots and continuous infusion of frusemide in cases of diuretic resistance, metolazone will be added for sequential blockade in the IV shots arm qualifying diuretic resistance, there will be second levle of randomization into time adjusted versus random time metolazone administration
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Frusemide IV shots = group A (Active Comparator): Frusemide as IV shots
  Interventions: Other: Frusemide IV shots
- Frusemide IV infusion = group B (Active Comparator): Frusemide as continuous IV infusion
  Interventions: Other: Frusemide IV infusion

INTERVENTIONS:
Other: Frusemide IV shots — giving frusemide by IV shots
  And if developed diuretic resistance (diminishing diuretic effect despite incremental dose of IV loop diuretic), adjuvant oral Metolazone will be given for sequential nephron blockade comparing its administration timed 60 minutes prior to the morning Frusemide shot versus given after. (This will be in a second level of randomization)
  Arms: Frusemide IV shots = group A
Other: Frusemide IV infusion — giving frusemide by continuous IV infusion
  And if developed diuretic resistance (diminishing diuretic effect despite incremental dose of IV loop diuretic), adjuvant oral Metolazone will be given for sequential nephron blockade
  Arms: Frusemide IV infusion = group B

SUMMARY:
1. Evaluate efficacy and safety of continuous infusion of IV Frusemide compared to IV shots in acute decompensated heart failure ADHF
2. Evaluate superiority of time-adjusted metolazone to morning frusemide IV shots compared to irrespective administration (at random times) to overcome diuretic resistance

DETAILED DESCRIPTION:
After admission for acute decompensated heart failure and ensuring eligibility to participate in the study, accepting patients will be randomized by a pre-prepared tables into 2 equal groups (A = shots, B = infusion): - Patients randomized to the Frusemide IV shots arm (group A) will be started on 80 mg frusemide daily (or at the least equal to their prior oral dose if was on >80 mg oral frusemide or equivalent doses of other loop diuretics). Dose will be allowed to be modified by judging the urine output in every 3 hours.

Patients randomized to continuous IV infusion arm (group B) will receive 84 mg Frusemide daily (40 mg bolus followed by 2 mg/ hour starting infusion rate). An extra bolus and/or modification of the infusion rate will be allowed after judging the urine output in 3 hours. The same regimen would be continued for at least 72 hours, or more than 72 hours if needed till switching to oral diuretics.

In patients who develop diuretic resistance defined as failure to achieve therapeutically desired urine output despite maximal doses of loop diuretics will be managed by adding thiazide type diuretic "Metolazone" to the regimen to achieve sequential nephron blockade. Metolazone (2.5 - 10 mg /day) addition will be allowed in both arms when deemed indicated, however, in the IV shots arm, there will be further 1:1 randomization for either giving metolazone timed 60 minutes before the morning IV frusemide shot (group A.T) or metolazone at random time irrespective of the frusemide dose timing (group A.R).

Variables that will be assessed in the patients to evaluate the prespecified end-points are:-

* Urine output in L/day as absolute volume and indexed volume to body weight.
* Weight loss in Kg as absolute number and in percentage of initial body weight.
* Diuretic efficiency defined as amount of urine output per 40mg frusemide.
* Impact on hemodynamics assessed by change in mean arterial pressure, inducing hypotension (systolic below 80 mmHg or requiring denovo vasopressors), or new clinical signs of hypoperfusion.
* Cumulative dose of IV frusemide per 72 hours.
* Improvement of NYHA class as judged by the treating physician.
* Number of days to introduction/restoring dose of betablockade therapy.
* Number of days to switch to oral diuretics as judged by the treating physician.
* Duration of ICU stay and of hospital stay.
* Change in serum creatinine (either rising or falling) in absolute value and percentage from baseline creatinine, as well as in eGFR equated by Cockcroft-Gold equation.
* Occurrence of worsening renal function (WRF) as defined by rise of serum creatinine by ≥ 0.3 mg/dl.
* Occurrence of 50% and or 100% rise in serum creatinine or indication to renal replacement therapy.
* Change in serum potassium as absolute value from baseline or below target range (between 4.0 - 5.0 mEq/dl). Serum potassium level will be routinely checked twice daily in the first 72 hours then once daily or every 48 hours as seen necessary.
* Inducing denovo hypomagnesemia (below 1.8mg/dl) or hyponatremia (below 135 mEq/dl)
* Rehospitalization within 30 days for new heart failure decompensation, and hospitalization for any cause.

VI. Study outcomes

1. Primary outcome

   * Time (in hours) to improvement of NYHA class when frusemide is given as shots compared to infusion.
   * Urine output (in ml/kg/h) per 40 mg of frusemide given as shots vs continuous infusion.
2. Secondary outcome(s)

   * Assessment of additive benefit of addition of metolazone to frusemide in ADHF.
   * Evaluating superiority of timely adjusted metolazone compared to given at random in overcoming resistance to IV frusemide (IV shots arm).

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years.
* Chronic heart failure prior diagnosis, based on signs and or symptoms of heart failure, presenting with acute decompensation as judged by the physician to require hospitalization for IV diuretics

Exclusion Criteria:

* Refusal to participate in the study.
* Allergy to IV frusemide.
* Severe renal impairment defined as eGFR<30ml/m.
* Cardiogenic shock or hemodynamic instability judged by the treating physician to be unsuitable to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-03-31 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Time to improvement of NYHA class | within 5 days
  Time (in hours) to improvement of NYHA class
Diuretic efficiency | 24 hours
  Urine output (in ml/kg/h) per 40 mg of frusemide given as shots vs continuous infusion.

SECONDARY OUTCOMES:
effectiveness of sequential nephron block | within 5 days of adding metolazone
  Assessing improvement of diuresis by adding of metolazone to frusemide in ADHF.patients who had developed diuretic resistance.
Evaluating superiority of timely adjusted metolazone compared to given at random in overcoming resistance to IV frusemide (only in IV shots arm) | within 5 days of adding metolazone
  Evaluating superiority of timely adjusted metolazone given 60 minutes prior to IV frusemide compared to when given at random in overcoming diuretic resistance (only in IV shots arm)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Shehata, MD, Study Chair — Cairo University; Magdy Abdelhamid, MD, Study Director — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Damman K, Testani JM. The kidney in heart failure: an update. Eur Heart J. 2015 Jun 14;36(23):1437-44. doi: 10.1093/eurheartj/ehv010. Epub 2015 Apr 2. PMID 25838436
- See also: Hoorn EJ, Ellison DH. Diuretic Resistance. Am J Kidney Dis. 2017;69(1):136-142. doi:10.1053/j.ajkd.2016.08.027 — https://linkinghub.elsevier.com/retrieve/pii/S027263861630511X